CLINICAL TRIAL: NCT03659604
Title: A Clustered Randomized Controlled Trial to Compare the Effectiveness of and Engagement in a Mobile Exergame 'SmartLife' With Tailored Feedback
Brief Title: Effectiveness of and Engagement in a Mobile Exergame With Tailored Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 'SmartLife' exergame
Record Dates: First submitted 2018-08-23; First posted 2018-09-06 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Physical Activity; Health Behavior
Keywords: physical activity; sedentary behavior; serious game; exergame; behaviour change techniques; tailored feedback
MeSH Terms: conditions — Motor Activity; Health Behavior; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Clustered randomized controlled trial/parallel assignment
  Different school classes will be allocated to one of the three groups: 1) intervention group with a game based on tailored feedback, 2) active control group with a game not using tailored feedback, 3) passive control group (waiting list group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental with tailored feedback (Experimental): 'SmartLife' with tailored feedback: School classes will receive the developed 'SmartLife' intervention with tailored feedback, that is based on data from a sensors that is integrated in a T-shirt.
  Interventions: Behavioral: 'SmartLife' with tailored feedback
- Active control without tailored feedback (Active Comparator): 'SmartLife' without tailored feedback: School classes will receive the developed 'SmartLife' intervention without tailored feedback.
  Interventions: Behavioral: 'SmartLife' without tailored feedback
- Passive control (Other): School classes will not receive any intervention, thus no game.
  Interventions: Behavioral: No game

INTERVENTIONS:
Behavioral: 'SmartLife' with tailored feedback — 'SmartLife' game with tailored feedback: mobile exergame with tailored feedback. Feedback will be based on accelerometer data from a sensor that is integrated in a T-shirt. The sensor captures individually calibrated accelerometer data and is paired with the mobile exergame. Depending on the physical activity intensity of the player, the game challenge and feedback adapts individually in real-time.
  Arms: Experimental with tailored feedback
Behavioral: 'SmartLife' without tailored feedback — 'SmartLife' without tailored feedback: mobile exergame without tailored feedback. The mobile exergame will not be paired to any sensor. The participant can play the mobile game, yet, will not receive any real-time feedback or adjustment in the game on physical activity intensity.
  Arms: Active control without tailored feedback
Behavioral: No game — Passive control: School classes will be asked to continue their daily life as usual.
  Arms: Passive control

SUMMARY:
The aim of this study is to investigate the effectiveness of the 'SmartLife' intervention on reducing sedentary behavior and increasing physical activity among adolescents and to investigate the engagement in the exergame. This will be compared in three groups: an intervention group that will receive a tailored exergame; an active control condition that will receive a non-tailored exergame; and a passive control condition that receives no intervention.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effectiveness of the 'SmartLife' intervention with tailored feedback on sedentary behavior and physical activity among adolescents and to investigate the engagement in the exergame. One intervention group will receive a version of the exergame that tailors feedback. This means tailored feedback will be based on data from a sensor which is integrated in a T-shirt and paired to the game. The active control group will receive a different version of the game, that does not provide tailored feedback.

Both groups will be compared to investigate their level of engagement in the game. A passive control group will be included that will be asked to continue their daily routines as usual. All three groups will be compared to determine the effectiveness of the 'SmartLife' intervention on physical activity and sedentary behavior.

ELIGIBILITY:
Inclusion Criteria:

* Between 12-18 years old
* Access to an Android smartphone (4.0.1) during study period
* No physical disabilities that hinder physical activity

Exclusion Criteria:

* Not Dutch-speaking
* Does not have access to an Android smartphone (4.0.1)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change in objectively measured physical activity (PA) | Baseline, 4 weeks, 8 weeks
  Change in amount of total physical activity and moderate-to-vigorous physical activity, measured via accelerometers

SECONDARY OUTCOMES:
Change in objectively measured sedentary behavior (SB) | Baseline, 4 weeks, 8 weeks
  Change in amount of total sitting time, measured via accelerometers
Change in subjectively measured Body Mass Index (BMI) | Baseline
  Change in BMI, measured via self-reported weight and height
Change in determinants of PA | Baseline, 4 weeks, 8 weeks
  Change in attitude, parental support, friends' co-participation, perceived social norm, self-efficacy, perceived benefits, perceived barriers, measured by validated items (questionnaire)
Change in determinants of SB | Baseline, 4 weeks, 8 weeks
  Change in attitude, self-efficacy, personal norm, social norm, social support of sedentary behavior (measured for the context of 1. TV viewing, game-play, and computer use), measured by validated items (questionnaire: correlates of context specific SB, Busschaert, 2015). Items are measured on a 5-point Likert scale (strongly disagree=1 - strongly agree=5). The average for each correlate will be calculated (meaning that sub scales for one correlate (e.g. attitude) will be combined).
Change in behavior of PA | Baseline, 4 weeks, 8 weeks
  Change in active transportation mode to school, measured by validated items (questionnaire: Flemish physical activity questionnaire, Verstaete et al., 2003), that measures the minutes engaged in different types of transportation to school. An average score for each component (walking, cycling, active transportation, passive transportation) will be calculated. Values will be indicated by minutes per day, whereby higher values will represent a better outcome, after reversing passive transportation.
Differences in engagement | 4 weeks
  Differences in engagement between intervention group and active control group, measured by validated items (questionnaire: Kids Game Experience Questionnaire), that measures immersion, narrative, pos/neg. affect, flow, absorption/involvement, transportation/immersion, challenge, tension/frustration. A scale ranges from 0 to 4, whereby higher values represent a better outcome. The average scores of the subscales represent each component, and a final averaged score for the GEQ questionnaire will be calcualted.
Differences in basic need satisfaction | 4 weeks
  Differences in basis need satisfaction between intervention group and active cotrol group, measured via 14 validated items (questionnaire)

OTHER OUTCOMES:
Location of engaging in PA | Baseline, 4 weeks, 8 weeks
  Location of engaging in PA, measured by validated items (questionnaire)
Differences usage of gameplay | 1 week, 2 weeks, 3 weeks, 4 weeks
  Differences in usage of game between intervention group and active controle group, measured via log data of the game (total number gameplay minutes) (log data)
Differences usage of game sessions | 1 week, 2 weeks, 3 weeks, 4 weeks
  Differences in usage of game between intervention group and active controle group, measured via log data of the game (total number gameplay sessions) (log data)
Differences usage of game in interaction with other players | 1 week, 2 weeks, 3 weeks, 4 weeks
  Differences in usage of game between intervention group and active controle group, measured via log data of the game (total number of interactions with other players) (log data)
Differences usage of game in invested game resources | 1 week, 2 weeks, 3 weeks, 4 weeks
  Differences in usage of game between intervention group and active controle group, measured via log data of the game (total number of invested game resources) (log data)
Differences usage of gameplay time | 1 week, 2 weeks, 3 weeks, 4 weeks
  Differences in usage of game between intervention group and active controle group, measured via log data of the game (gameplay time: measured via 1-3, indicating morning, afternoon, evening) (log data)
Differences usage of gameplay location | 1 week, 2 weeks, 3 weeks, 4 weeks
  Differences in usage of game between intervention group and active controle group, measured via log data of the game (gameplay location, indicating 1-2; 1=inside/2=outside) (log data)
Usage of game physical activity | 1 week, 2 weeks, 3 weeks, 4 weeks
  Usage of game by intervention group, measured via log data of the game (average moderate to vigorous physical activity) (log data)
Usage of game sedentary behaviour | 1 week, 2 weeks, 3 weeks, 4 weeks
  Usage of game by intervention group, measured via log data of the game (sedentary behaviour) (log data)

CONTACTS AND LOCATIONS:
Overall Officials: Greet Cardon, Professor, Principal Investigator — University Ghent; Ann DeSmet, Dr., Principal Investigator — University Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No